CLINICAL TRIAL: NCT03184012
Title: Clinical Comparison Between Zirconia Crowns Versus Anterior Strip Crowns
Brief Title: Clinical Evaluation of Zirconia Crowns and Anterior Strip Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Bashaer S. Abdulhadi, Dr. Bashaer Abdulhadi, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: King Abdulaziz University
Record Dates: First submitted 2017-06-02; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Dental Caries
Keywords: caries; full coverage; strip crown; Zirconia crown; primary anterior teeth; crown
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: one group assigned to be treated with Zirconia crowns, the other group assigned to be treated with resin composite strip crowns
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NuSmile Zirconia crowns (Experimental): NuSmile Zirconia crowns is an esthetic primary anterior crown used to restore carious primary anterior teeth.
  Interventions: Device: NuSmile Zirconia crowns by NuSmile company
- Composite resin strip crowns (Experimental): Composite resin strip crowns is an esthetic conventional primary anterior crown used to restore carious primary anterior teeth.
  Interventions: Device: Composite resin strip crowns by 3M company

INTERVENTIONS:
Device: NuSmile Zirconia crowns by NuSmile company — anterior carious teeth restored with Zirconia crowns
  Arms: NuSmile Zirconia crowns
Device: Composite resin strip crowns by 3M company — anterior carious teeth restored with Strip crowns
  Arms: Composite resin strip crowns

SUMMARY:
The hypothesis to be investigated is that no difference will be found upon comparing resin composite strip crowns and NuSmile zirconia crowns (NuSmile ZR) esthetic primary anterior in restoring anterior primary teeth.

DETAILED DESCRIPTION:
The aim of this study is to clinically evaluate the performance of a new NuSmile ZR esthetic primary anterior crowns, compared with anterior resin composite strip crowns in the restoration of 120 teeth (primary incisors and lateral anterior teeth in the deciduous dentition of child patients).

ELIGIBILITY:
Inclusion Criteria:

* Healthy Children with no history of any systemic illness or any developmental disease of the teeth and jaws that would have affected dietary patterns, caries, susceptibility or the selection of restorative materials to the best of current knowledge.
* Minimal of two surfaces of caries in the targeted tooth.
* Patient with Early Childhood Caries as defined by American Academy of Pediatric Dentistry (AAPD), 2016.
* Cooperative patient who had behavioral rating "positive" or "definitely positive" followed the Frankl behavior classification scale. (Frankl et al. 1962)
* Opposing teeth present.
* Written consent was obtained from the parent/guardian after explaining the full details of the treatment procedure and its possible outcomes, discomfort, risks, and benefits.
* No patient was excluded on the basis of gender, race, social or economic background.

Exclusion Criteria:

* Teeth with proximity to exfoliation and resorption of the root passed its half.
* Patients with allergy or hypersensitivity to nickel in case of posterior group teeth.
* Presence of single surface caries not involving the proximal surfaces.
* Teeth that has been subjected to trauma.
* Anxious, uncooperative patients who need to be treated under general anesthesia.
* Children who suffer from bruxism.
* Children with special needs.
* Presence of tooth wear on the opposing teeth (in case of anterior teeth), or absence of opposing.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Gingival Health | 3-month follow-up
  This parameter was evaluated using a blunt periodontal probe (Double ended probe Williams 1-2-3-5-7-8-9-10 Goldman Fox Flat) according to the Löe and Silness gingival index [Löe, 1967].
Plaque index | 3-month follow-up
  This parameter was evaluated using a blunt periodontal probe (Double ended probe Williams 1-2-3-5-7-8-9-10 Goldman Fox Flat) according to the Löe and Silness gingival index [Löe,1967].
Restoration failure | 3-month follow-up
  This was clinically evaluated with visual assessment of the restoration, according to the US Public Health Service "USPHS", Alpha criteria rating system [Ryge, 1980].
Tooth wear of opposing dentition | 3-month follow-up
  Tooth wear was evaluated according to the Smith and Knight Tooth Wear Index (Bardsley, 2008; Smith and Knight, 1984)
Gingival Health | 6-month follow-up
  This parameter was evaluated using a blunt periodontal probe (Double ended probe Williams 1-2-3-5-7-8-9-10 Goldman Fox Flat) according to the Löe and Silness gingival index [Löe, 1967].
Plaque index | 6-month follow-up
  This parameter was evaluated using a blunt periodontal probe (Double ended probe Williams 1-2-3-5-7-8-9-10 Goldman Fox Flat) according to the Löe and Silness gingival index [Löe, 1967].
Restoration failure | 6-month follow-up
  This was clinically evaluated with visual assessment of the restoration, according to the US Public Health Service "USPHS", Alpha criteria rating system [Ryge, 1980].
Tooth wear of opposing dentition | 6-month follow-up
  Tooth wear was evaluated according to the Smith and Knight Tooth Wear Index (Bardsley, 2008; Smith and Knight, 1984)
Gingival Health | 12-month follow-up
  This parameter was evaluated using a blunt periodontal probe (Double ended probe Williams 1-2-3-5-7-8-9-10 Goldman Fox Flat) according to the Löe and Silness gingival index [Löe, 1967].
Plaque index | 12-month follow-up
  This parameter was evaluated using a blunt periodontal probe (Double ended probe Williams 1-2-3-5-7-8-9-10 Goldman Fox Flat) according to the Löe and Silness gingival index [Löe, 1967].
Restoration failure | 12-month follow-up
  This was clinically evaluated with visual assessment of the restoration, according to the US Public Health Service "USPHS", Alpha criteria rating system [Ryge, 1980].
Tooth wear of opposing dentition | 12-month follow-up
  Tooth wear was evaluated according to the Smith and Knight Tooth Wear Index (Bardsley, 2008; Smith and Knight, 1984)

CONTACTS AND LOCATIONS:
Overall Officials: Bashaer S Abdulhadi, MSc, Principal Investigator — King Abdulaziz University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alaki SM, Abdulhadi BS, AbdElBaki MA, Alamoudi NM. Comparing zirconia to anterior strip crowns in primary anterior teeth in children: a randomized clinical trial. BMC Oral Health. 2020 Nov 10;20(1):313. doi: 10.1186/s12903-020-01305-1. PMID 33167954